CLINICAL TRIAL: NCT04229069
Title: Randomized, Double-blind, Placebo-controlled Intervention Study on Effects of Basica® on Acid-base Balance, Metabolism and Quality of Life in Elderly Healthy Volunteers.
Brief Title: Acid-Base Balance, Metabolism and Minerals
Acronym: BASICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Boschmann, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASICA
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Acid-Base Balance Disorder; Metabolic Acidosis
Keywords: acid-base balance; energy metabolism; protein-rich diet; alkaline supplementation; calorimetry; microdialysis; randomized placebo-controlled trial
MeSH Terms: conditions — Acidosis | interventions — basica

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basica (Active Comparator): 4-week dietary supplementation with an alkaline salt (Basica)
  Interventions: Dietary Supplement: alkaline salt mixture
- Placebo (Placebo Comparator): 4-week dietary supplementation with a placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: alkaline salt mixture — blood and tissue alkalinisation
  Other Names: Basica
  Arms: Basica
Dietary Supplement: placebo — no blood and tissue alkalinisation
  Arms: Placebo

SUMMARY:
Metabolism is controlled by macro- and micronutrients. Protein-rich diets should lead to latent acidosis at tissue level with further negative implications. Food supplements with alkaline salts are available and popular pretending to prevent these changes.

Within a randomized double-blind placebo-controlled trial, the investigators tested the hypotheses 1) that a 4-week protein-rich diet induces a latent tissue acidosis and 2) an alkaline supplement can compensate this. Acid-base balance and important metabolic parameters were determined before and after 4 weeks of supplementation by peripheral blood samples, indirect calorimetry and muscle microdialysis before and after a protein-rich test meal.

ELIGIBILITY:
Inclusion Criteria:

* slightly reduced kidney function (GFR 60-89 ml/min)
* Body mass index 20.0 - 29.9 kg/m2
* normal daily diet composition: 45-50, 35-40, and 15 E% from carbs, fats and proteins, respectively

Exclusion Criteria:

* sorbitol-/fructose-intolerance
* intake of antacidic drugs
* vegetarians, vegans
* intake of any nutritional supplements
* any cardiovascular, pulmonary, endocrine or metabolic diseases
* any drug abuse
* intake of any anticoagulant drugs

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle dialysate lactate-pyruvate ratio | before and after 4-weeks of supplementation at baseline (after a 12 hours overnight fast) and 60, 120, and 180 minutes after a protein-enriched test meal
  surrogate measure for muscle tissue pH

IPD SHARING:
Plan to Share IPD: No